CLINICAL TRIAL: NCT02649920
Title: Pilot, Comparative, Not Randomized, Two Centers Study Comparing the Efficiency of Cervical Ripening BALLoon (Cook) to the DINOprostone (Propess) for the Cervical Maturation in Case of Unfavorable Cervix (Bishop <6) in the Population of Obese Pregnant Women (BMI >= 30 kg/m²)
Brief Title: Comparing the Efficiency of Cervical Ripening BALLoon (Cook) to the DINOprostone (Propess) for the Cervical Maturation in Case of Unfavorable Cervix (Bishop <6) in the Population of Obese Pregnant Women (BMI >= 30 kg/m²)
Acronym: BALLODINO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed inclusion
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD019-15
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Delivery
Keywords: unfavorable cervix; obese pregnant women
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical ripening balloon (Experimental): Prospective
  Interventions: Device: Cervical ripening balloon
- Dinoprostone (Active Comparator): Retrospective
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Device: Cervical ripening balloon
  Other Names: Cook
  Arms: Cervical ripening balloon
Drug: Dinoprostone
  Other Names: Propess
  Arms: Dinoprostone

SUMMARY:
At the moment in France, one delivery on four is induced for a medical indication. In this context, the practitioners are exposed to an additional difficulty when the clinical examination of the patient reveals a unfavorable cervix because the main drug used for the releases cannot be used and the cervix must be previously mature.

There is a pharmacological method used and estimated in these indications of cervical maturation: the dinoprostone (Propess®).

Other methods using a mechanical process, are under development and of evaluation as it is the case of the probe of dilation with double balloon (Cook®).

The population of the obese women is a population in constant increase in France and presenting deliveries to higher risks of maternal and foetal complications. At these patients, the medicinal releases seem also more difficult and at greater risks of failures.

The investigators wish compared the efficiency of the cervical ripening balloon to the dinoprostone within the framework of a medical indication in a release with a unfavorable cervix in obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Term ≥ 37 weeks of amenorrhea
* Singleton pregnancy
* Cephalic presentation
* Medical indication of release and unfavorable cervix (Bishop <6)
* BM pre-pregnancy ≥ 30 kg/m2
* Having given their agreement for the participation of the study
* Patient receiving social coverage

Exclusion Criteria:

* Age < 18 years
* Term < 37 weeks of amenorrhea
* Multiple pregnancy
* Favorable cervix (Bishop ≥ 6)
* Contraindication of vaginal delivery: praevia placenta, transverse presentation, cord prolapse
* Evolutive urinary tract infection (positive urine dip: leukocytes/ nitrites)
* Not affiliated with a legal protection regime
* Patient trust, guardianship, under legal protection measure, deprived of freedom

Balloon's contraindications:

* Abnormal pelvis structure
* Evolutive genital herpes
* Invasive cervical cancer
* Anomaly of foetal heart rate
* Breech presentation
* Maternal heart disorder
* Hydramnios
* Serious and uncontrolled arterial high blood pressure
* Rupture of membranes
* Medical histories of hysterotomy, classic uterine section, myomectomy or quite different uterine section of full thickness
* Presentation above superior pelvic strait

Dinoprostone's contraindications:

* Scarred uterus
* Prostaglandin's hypersensitivity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, PH, Study Director — Centre Hospitalier Departemental Vendee
Locations (2):
- France (2):
  - Centre Hospitalier Vendée, La Roche-sur-Yon
  - Centre Hospitalier, Le Mans

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Ripening Balloon: Prospective
  Cervical ripening balloon
- Dinoprostone: Retrospective
  Dinoprostone
Period: Overall Study
Arm/Group | Cervical Ripening Balloon | Dinoprostone
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The sponsor took the decision to stop the inclusions prematurely as of 23/11/2016. No statistical analysis was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Ripening Balloon | Dinoprostone | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — The sponsor took the decision to stop the inclusions prematurely as of 23/11/2016. No statistical analysis was performed.
  years | 26.5 (2.12) |  | 26.5 (2.12)
Sex: Female, Male [Count of Participants; unit: Participants] — The sponsor took the decision to stop the inclusions prematurely as of 23/11/2016. No statistical analysis was performed.
  Participants
    Female | 2 |  | 2
    Male | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Bishop Score After 24 Hours of Maturation
Time Frame: 24 hours
Population: Data were not collected.
Arm/Group | Cervical Ripening Balloon | Dinoprostone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Death, serious adverse event and other (non serious adverse event) were not assessed for the study
Arm/Group | Cervical Ripening Balloon | Dinoprostone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No